CLINICAL TRIAL: NCT05153317
Title: A Phase 3 Open-label Study Evaluating the Long-term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor Triple Combination Therapy in Cystic Fibrosis Subjects 2 Years and Older
Brief Title: Evaluation of Long-term Safety and Efficacy of ELX/TEZ/IVA in Cystic Fibrosis (CF) Participants 2 Years and Older
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX20-445-112; 2020-002239-31 (EudraCT Number)
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX/TEZ/IVA (Experimental): Participants will receive ELX/TEZ/IVA in the morning and IVA in the evening.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination granules or tablets for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Granules or tablets for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
The purpose of this study is to evaluate the long term safety, tolerability, efficacy and pharmacodynamics of elexacaftor (ELX)/tezacaftor (TEZ)/ivacaftor (IVA) in CF participants 2 years of age and older.

ELIGIBILITY:
key Inclusion Criteria:

* Completed study drug treatment in the parent study (VX20-445-111 Part B, NCT04537793), or had study drug interruption(s) in the parent study, but did not permanently discontinue study drug, and completed study visits up to the last scheduled visit of the Treatment Period of the parent study

Key Exclusion Criteria:

* History of study drug intolerance in the parent study
* History of poor compliance with ELX/TEZ/IVA and/or procedures in the parent study

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Week 196

SECONDARY OUTCOMES:
Absolute Change in Sweat Chloride (SwCl) | From Baseline up to Week 192
Absolute Change in Lung Clearance Index (LCI) 2.5 | From Baseline up to Week 192

CONTACTS AND LOCATIONS:
Locations (22):
- United States (13):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - NC TraCS Institute - CTRC University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Telethon Kids Institute, Nedlands
  - The Royal Children's Hospital, Parkville
  - Queensland Children's Hospital, South Brisbane
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- Germany (2):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitatsklinikum Essen (AoR), Kinderklinik III, Abt. fur Pneumologie, Essen
- United Kingdom (2):
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing